CLINICAL TRIAL: NCT00233454
Title: A Single Arm, Phase 2, Open-Label Study to Determine the Efficacy of Twice Daily Oral Dosing of PKC412 <Midostaurin> Administered to Patients With Aggressive Systemic Mastocytosis (ASM) and Mast Cell Leukemia (MCL)
Brief Title: Phase 2 Midostaurin in Aggressive Systemic Mastocytosis and Mast Cell Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jason Robert Gotlib (Other)
Collaborators: Novartis (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Jason Robert Gotlib, Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-13704; 95242 (Other: Stanford University Secondary IRB Approval Number); HEMMPD0003 (Other: OnCore); CPKC412D2201 (Other: Novartis, Inc); 2213 (Other: Novartis, Inc)
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Results first posted 2015-07-09 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Systemic Mastocytosis, Aggressive (ASM); Leukemia, Mast Cell; Hematological Non-mast Cell Lineage Disease (AHNMD)
MeSH Terms: conditions — Mastocytosis, Systemic; Aggression; Leukemia, Mast-Cell | interventions — midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Midostaurin (Experimental): 100 mg midostaurin twice daily as oral capsules
  Interventions: Drug: Midostaurin

INTERVENTIONS:
Drug: Midostaurin — Midostaurin is a broad-spectrum protein kinase inhibitor, acting on conventional PKC isoforms (α, β, γ); PDFRβ; VEGFR2; Syk; PKCη; Flk-1; Flt3; Cdk1/B; PKA; c-Kit; c-Fgr; c-Src; VEGFR1; and EGFR
  Other Names: PKC412; CGP41251; CGP41231

SUMMARY:
The safety and efficacy of midostaurin (PKC412), a novel investigational drug, will be evaluated on the basis of response rate, when administered to patients with aggressive systemic mastocytosis (ASM) or mast cell leukemia (MCL)

DETAILED DESCRIPTION:
This study assesses the activity and safety profile of twice-daily oral doses of midostaurin in patients with aggressive systemic mastocytosis (ASM) or mast cell leukemia (MCL) with or without associated clonal hematological non-mast cell lineage disease (AHNMD).

Aggressive systemic mastocytosis (ASM) and mast cell leukemia (MCL) are characterized by excessive bone marrow production of mast cells which can can infiltrate tissues and release harmful substances, resulting in organ damage. These diseases have very limited treatment options and poor prognosis. Existing treatments for in advanced mast cell disease, eg, interferon-alpha; corticosteroids; and/or cladribine, exhibit low response rates that are usually partial in nature.

ELIGIBILITY:
Inclusion criteria

* At least 18 years of age.
* Karnofsky performance status (KPS) of > 30% (equivalent to ECOG 0 to 3)
* Mast cell disease, histologically confirmed and documented to be

  * Aggressive systemic mastocytosis (ASM) OR
  * Mast cell leukemia (MCL) meeting the following criteria

    * Meets criteria for systemic mastocytosis
    * Biopsy indicates diffuse infiltration by atypical, immature mast cells
    * Bone marrow aspirate smears show at least 20% mast cells
* Confirmed availability of tissue sample within 6 months prior to entry into study, for evaluation of KIT mutation status of the tumor cells. Subjects who have systemic mastocytosis PLUS eosinophilia AND known positivity for FIP1L1-PDGFR-alpha fusion are eligible only if they have demonstrated relapse or disease progression on prior imatinib therapy
* Blood levels of liver enzymes within normal limits (EXCEPTION: If the sole cause of elevated blood levels of liver enzymes is ASM/MCL, then AST and ALT ≤ 4X upper limit of normal (ULN), and/or bilirubin ≤ 4X ULN)
* Serum creatinine < 2.0 mg/dL
* If ANC < 1500/mm3; Hb < 10 g/dL; platelets < 75,000/mm3; AND/OR other blood values are > grade 2, then the relationship of these cytopenia(s) should be established as related to ASM or MCL on the basis of presence of mast cell infiltrate in the screening bone marrow exam and/or the presence of disease-related hypersplenism
* Prior use of glucocorticoids must be tapered off within 14 days of Day 1 of midostaurin treatment (EXCEPTION: If in the opinion of the investigator, the subject can be tapered off glucocorticoids, then dosage should be tapered to the minimal dose possible before first treatment with midostaurin)
* Negative serum pregnancy test for women of childbearing potential within 48 hours prior to administration of study drug
* Written informed consent.
* Anyone of reproductive potential must agree to use barrier contraceptives for the duration of the study
* Women of childbearing potential must have a negative serum pregnancy test 48 hours prior to administration of study drug, and must agree to:

  * Use barrier contraception for the duration of the study
  * Use barrier contraception for 3 months post-study
  * Not breast-feed

Exclusion criteria

* Active pulmonary disease based on physical assessment or lateral chest X-ray, considered by the investigator to be unrelated to mastocytosis
* Any pulmonary infiltrate or abnormality on the baseline chest X-ray known to be new in the previous 4 weeks (EXCEPTION: pleural effusion related to systemic mastocytosis, eg, secondary to ascites, AND not causing symptomatic respiratory complaints, may be eligible)
* Cardiovascular disease, including congestive heart failure
* Myocardial infarction within 6 months
* Poorly-controlled hypertension with any Grade 3/4 cardiac problems (per New York Heart Association Criteria)
* Uncontrolled diabetes
* Chronic renal disease
* Active uncontrolled infection
* Known malignant disease involving the central nervous system (CNS)
* Known confirmed diagnosis of HIV infection or active viral hepatitis.
* Any other known disease, or concurrent severe and/or uncontrolled medical condition which could compromise participation in the study, including but not limited to:
* Received any investigational agent, chemotherapy, or 2-chlorodeoxyadenosine (2-CdA) within 30 days prior to Day 1 of PKC412 treatment.
* Received interferon-alpha within 30 days prior to Day 1 of midostaurin treatment.
* Received hematopoietic growth factor support within 14 days of Day 1 of midostaurin treatment.
* Any surgical procedure, excluding central venous catheter placement or other minor procedures (eg, skin biopsy) within 14 days of Day 1 of midostaurin treatment
* Pregnant or breast-feeding
* Unwilling or unable to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2005-03 (Actual); Primary Completion 2010-06-18 (Actual); Study Completion 2011-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Robert Gotlib, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Stanford University School of Medicine, Stanford, California
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University-St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paschka P, Marcucci G, Ruppert AS, Mrozek K, Chen H, Kittles RA, Vukosavljevic T, Perrotti D, Vardiman JW, Carroll AJ, Kolitz JE, Larson RA, Bloomfield CD; Cancer and Leukemia Group B. Adverse prognostic significance of KIT mutations in adult acute myeloid leukemia with inv(16) and t(8;21): a Cancer and Leukemia Group B Study. J Clin Oncol. 2006 Aug 20;24(24):3904-11. doi: 10.1200/JCO.2006.06.9500. PMID 16921041
- [Result] Gotlib JR, George TI, Linder A, et al. "Phase II Trial of the Tyrosine Kinase Inhibitor PKC412 in Advanced Systemic Mastocytosis: Preliminary Results." Blood. 16 November 2006;108(11)16:abs3609
- [Result] Gotlib JR, George TI, Corless C, et al. "The KIT Tyrosine Kinase Inhibitor Midostaurin (PKC412) Exhibits a High Response Rate in Aggressive Systemic Mastocytosis(ASM): Interim Results of a Phase 2 Trial." Blood. 16 November 2007;110(11):abs 3536
- [Result] Gotlib JR, DeAngelo DJ, George TI, et al. "KIT Inhibitor Midostaurin Exhibits a High Rate of Clinically Meaningful and Durable Responses in Advanced Systemic Mastocytosis: Report of a Fully Accrued Phase II Trial." Blood. 19 November 2010;116(21):abs316
- [Result] Gotlib J, Kluin-Nelemans HC, George TI, Akin C, Sotlar K, Hermine O, Awan FT, Hexner E, Mauro MJ, Sternberg DW, Villeneuve M, Huntsman Labed A, Stanek EJ, Hartmann K, Horny HP, Valent P, Reiter A. Efficacy and Safety of Midostaurin in Advanced Systemic Mastocytosis. N Engl J Med. 2016 Jun 30;374(26):2530-41. doi: 10.1056/NEJMoa1513098. PMID 27355533
- [Result] DeAngelo DJ, George TI, Linder A, Langford C, Perkins C, Ma J, Westervelt P, Merker JD, Berube C, Coutre S, Liedtke M, Medeiros B, Sternberg D, Dutreix C, Ruffie PA, Corless C, Graubert TJ, Gotlib J. Efficacy and safety of midostaurin in patients with advanced systemic mastocytosis: 10-year median follow-up of a phase II trial. Leukemia. 2018 Feb;32(2):470-478. doi: 10.1038/leu.2017.234. Epub 2017 Jul 24. PMID 28744009

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Midostaurin
Started | 26
2 Months (for Response Rate) | 26
Completed | 20
Not Completed | 6
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Arm/Group | Midostaurin
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 13
Age, Continuous [Median (Full Range); unit: years] | 65 [24.8 to 79.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26
Disease Sub-type [Count of Participants; unit: Participants] — Systemic mastocytosis (SM) is comprised of 3 primary sub-types, aggressive SM (ASM); SM with an associated hematologic neoplasm (SM-AHN); and mast cell leukemia (MCL).
  Participants
    Aggressive systemic mastocytosis (ASM) | 3
    SM with associated hematologic neoplasm (SM-AHN) | 17
    Mast cell leukemia (MCL) | 6

OUTCOME MEASURES:

1. Primary Outcome: Subjects With Clinical Response [Partial Response (PR) + Complete Response (CR)]
Description: Clinical Response [PR + CR] will be assessed after 2 cycles of treatment, with each cycle being 28 days (4 weeks) in length.
  Except as otherwise noted, the minimum criteria for PR is improvement by at least 50% from the baseline value towards the indicated value for one or more of the criteria below:
  BONE MARROW & BLOOD
  * ANC <1000/uL
  * Hb <10 g/dL
  * Platelets >100,000/uL LIVER
  * If hepatomegaly with ascites, decrease in frequency of paracenteses by 50%
  * Elevated enzyme levels > upper limit of normal (ULN)
  * Hypoalbuminemia < ULN
  * Portal hypertension > ULN SPLEEN
  * If palpable splenomegaly with hypersplenism/thrombocytopenia, hypersplenism markers improved GI TRACT
  * If malabsorption with hypoalbuminemia and/or weight loss, albumin improved BONES
  * If huge osteolyses or/and severe osteoporosis with pathologic fractures, partial resolution of osteolyses
  Subjects with PR or greater continue, those without response discontinue.
Time Frame: 2 months
Measure: Number; unit: participants
Arm/Group | Midostaurin
Number analyzed (Participants) | 26
participants | 25

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival will be assessed after 12 cycles of treatment, with each cycle being 28 days (4 weeks) in length. 12 cycles of treatment is considered to be about 11 months.
Time Frame: 11 months
Measure: Number; unit: participants
Arm/Group | Midostaurin
Number analyzed (Participants) | 26
participants | 20

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was assessed as the median duration of survival at the time of data cut-off, and reported with 95% confidence interval.
Time Frame: 40 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Midostaurin
Number analyzed (Participants) | 26
months | 40 [27.3 to 52.7]

ADVERSE EVENTS:
Time Frame: This study includes open-ended maintenance treatment. AEs are reported for the duration of treatment through follow-up to death or lost-to-follow-up.
Arm/Group | Midostaurin
All-Cause Mortality (participants affected / at risk) | 7/26
Serious Adverse Events (participants affected / at risk) | 12/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midostaurin (N=26)
Blood and lymphatic system disorders - Other, hand swelling (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (5)
vomiting (Gastrointestinal disorders) | 1 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (3)
Dehydration (Gastrointestinal disorders) | 1 (3)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Death NOS-refactory sepsis (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
General disorders - Other, increased fatigue with "cloudy thinkin (General disorders) | 1 (3)
Hepatobiliary disorders - Other, Liver lesions-neuroendocrine tumor (Hepatobiliary disorders) | 1 (1)
Infections and infestations - Other, Urosepsis (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (3)
Scrotal infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (2)
Nervous system disorders - Other, transient ischemic attack/ cerebrovascular accident (Nervous system disorders) | 1 (1)
Renal and urinary disorders - Other, Hematuria (Renal and urinary disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, blistery lesions on hands and lower arms (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midostaurin (N=26)
Anemia (Blood and lymphatic system disorders) | 11 (12)
Blood and lymphatic system disorders - Other, lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (5)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Blurred vision (Eye disorders) | 3 (3)
Cataract (Eye disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Ascites (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 12 (12)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Enterocolitis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other, increased saliva (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, bowel obstruction (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 24 (24)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 18 (18)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 9 (9)
Fatigue (General disorders) | 13 (14)
Fever (General disorders) | 6 (6)
Flu like symptoms (General disorders) | 4 (4)
Gait disturbance (General disorders) | 2 (2)
General disorders and administration site conditions - Other, altitude sickness (General disorders) | 1 (1)
General disorders and administration site conditions - Other, failure to thrive (General disorders) | 1 (1)
General disorders and administration site conditions - Other, fluid retention (General disorders) | 1 (1)
General disorders and administration site conditions - Other, malnutrition (General disorders) | 1 (1)
General disorders and administration site conditions - Other, transfusion reaction (General disorders) | 1 (1)
General disorders and administration site conditions - Other, weakness (General disorders) | 3 (3)
General disorders and administration site conditions - Other, thrush (General disorders) | 1 (1)
General disorders and administration site conditions - Other animal or insect bite (General disorders) | 3 (3)
Localized edema (General disorders) | 2 (2)
Pain (General disorders) | 3 (5)
Hepatobiliary disorders - Other, increased Hepatosplenomegaly (Hepatobiliary disorders) | 5 (5)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Infections and infestations - Other, (tooth, peritoneal catheter) (Infections and infestations) | 2 (2)
Infections and infestations - Other, herpes lesion(nasal/oral) (Infections and infestations) | 3 (3)
Infections and infestations - Other, herpes zoster (Infections and infestations) | 1 (1)
Infections and infestations - Other, Lyme's disease (Infections and infestations) | 1 (1)
Infections and infestations - Other, peritonitis (Infections and infestations) | 1 (1)
Infections and infestations - Other, skin (cellulitis) (Infections and infestations) | 2 (2)
Infections and infestations - Other, staph infection (Infections and infestations) | 2 (2)
Infections and infestations - Other, Urosepsis (Infections and infestations) | 1 (1)
Infections and infestations - Other, viral (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (2)
Creatinine increased (Investigations) | 3 (3)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (2)
Investigations - Other, tryptase increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 6 (9)
Platelet count decreased (Investigations) | 8 (8)
Weight gain (Investigations) | 4 (5)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 2 (3)
Serum Amylase Increased (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (7)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, rotator cuff tear (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, basal cell CA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, squamous cell CA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Treatment related secondary malignancy, lung CA, malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 8 (8)
Nervous system disorders - Other, lightheadedness (Nervous system disorders) | 6 (6)
Nervous system disorders - Other, presyncope (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, vertigo (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 4 (4)
Confusion (Psychiatric disorders) | 4 (4)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3)
Psychosis (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Skin and subcutaneous tissue disorders - Other, dermatitis (blisters) (Skin and subcutaneous tissue disorders) | 4 (4)
Skin and subcutaneous tissue disorders - Other, injury (abrasion) (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, not specified (Skin and subcutaneous tissue disorders) | 2 (3)
Skin and subcutaneous tissue disorders - Other, skin nodule (Skin and subcutaneous tissue disorders) | 2 (3)
Skin and subcutaneous tissue disorders - Other, sunburn (Skin and subcutaneous tissue disorders) | 2 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 4 (4)
Hematoma (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 2 (2)
Vascular disorders - Other, conjunctival hemorrhage (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No